CLINICAL TRIAL: NCT02478710
Title: Aerosolized Antibiotics in the Treatment of Ventilator Associated Pneumonia: A Pilot Study
Brief Title: Aerosolized Antibiotics in the Treatment of Ventilator Associated Pneumonia
Acronym: AAINTVAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6517
Record Dates: First submitted 2015-04-30; First posted 2015-06-23 (Estimated); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Vancomycin; Tobramycin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerosolized Placebo (Placebo Comparator): Placebo tobramycin 0.5 mL 0.9% normal saline q.12h. Placebo vancomycin 0.5 mL 0.9% normal saline q.8h.
  Interventions: Drug: Aerosolized Placebo
- Aerosolized Tobramycin or Vancomycin (Experimental): Aerosolized tobramycin 300 mg diluted in 5 mL 0.9% normal saline q.12h. Aerosolized vancomycin 125 mg diluted in 5 mL 0.9% normal saline q.8h.
  Interventions: Drug: Aerosolized Tobramycin or Vancomycin

INTERVENTIONS:
Drug: Aerosolized Tobramycin or Vancomycin — Tobramycin: 300 mg diluted in 5 mL of 0.9% normal saline q.12h. Vancomycin: 125 mg diluted in 5 mL 0.9% normal saline q.8h.
  Other Names: Tobi, Tobrex; Vancocin
  Arms: Aerosolized Tobramycin or Vancomycin
Drug: Aerosolized Placebo — Placebo tobramycin: 5 ml 0.9% normal saline q. 12h. Placebo vancomycin: 5m 0.9% normal saline q. 8 hr.
  Other Names: Normal saline solution
  Arms: Aerosolized Placebo

SUMMARY:
The purpose of this study is to determine if administering inhaled antibiotics directly into the lungs in conjunction with intravenous (IV) antibiotics leads to better outcomes and decreased recurrence of ventilator associated pneumonia (VAP) when compared to IV antibiotics alone.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) remains a serious problem in critically ill patients with an incidence of 8-28% and mortality ranging from 24-57%. A landmark study comparing eight days versus fifteen days of antibiotic therapy reported a pulmonary infection recurrence rate of 26-29%. Costs associated with VAP can reach up to $40,000 per occurrence.

Aerosolized antibiotics have been used to treat ailments such as cystic fibrosis and bronchiectasis. Previous research indicates that aerosolized antibiotics attain a 200 fold greater concentration in the lung than in the blood, and that sputum trough levels remain 20 fold greater than that of acceptable serum antibiotic troughs. Additionally, aerosolized antibiotics are considered safe (without increased risk of bacterial resistance) with better treatment success when compared to controls (OR 2.75, 95% CI 1.06-7.17), although no mortality benefit has been identified. Some studies have shown reduced systemic toxicity when using aerosolized antibiotics while others have shown no difference. Aerosolized tobramycin prevents pseudomonas infections in patients with Cystic Fibrosis. Furthermore aerosolized antibiotics improve pulmonary function in these patients, including Forced Expiratory Volume in 1 second (FEV1), and decrease the need for hospitalization. Lung transplant patients and patients with Human Immunodeficiency Virus (HIV) also benefit from aerosolized fungal prophylaxis and treatment. The benefit has been less clear in patients with non-Cystic Fibrosis bronchiectasis, and although some studies show benefits to aerosolized antibiotics in preventing and treating nosocomial pneumonias, no large prospective randomized trials have been performed to confirm the benefit or to change practice recommendations.

Antimicrobials must reach the site of infection, bind the target site, and remain bound for a sufficient time period to disrupt the life cycle of the cells. Only 21% of an administered antibiotic dose actually ends up in the lung parenchyma. Multiple studies have shown that the ideal particle size for inhalation is between 1 and 5 microns. Particles that are too small get exhaled, and particles that are too large do not reach the alveoli. Non-humidified nebulization is better for drug administration than humidified air. Isotonicity of the drug, pH, and the presence of preservatives in the solution also need to be evaluated for optimal drug delivery and function. The ideal method of administration of aerosolized antibiotics also remains to be determined.

Inhaled tobramycin has been used in several studies over the past thirty years, mostly in patients with Cystic Fibrosis. It has been shown to be effective in decreasing sputum colony counts of Pseudomonas Aeruginosa. Inhaled gentamycin has also been shown to delay acquisition of Pseudomonas in children with Cystic Fibrosis, as well as decreasing disease progression. Chest tightness and persistent cough are the side effects mentioned within these studies. This suggests that inhalation is a safe method for the administration of tobramycin.

It has been shown that in Community-Acquired Pneumonia (CAP) the alveolar macrophages initiate a pro-inflammatory cascade. Failure to control excessive inflammation, leads to an exaggerated systemic response resulting in organ damage. Local and systemic levels of these pro-inflammatory mediators have been shown to correlate with the severity of disease. The investigators speculate that a similar response exists in patients with VAP.

The investigators propose a prospective, randomized trial designed to assess the value of aerosolized antibiotics in the treatment of ventilator associated pneumonia and to evaluate the impact of co-existing, non-bacterial pathogens and cytokines on the ability to clear pneumonia in culture-proven cases of VAP. Eligible patients will be randomized at the time of bronchoalveolar lavage or combicath to receive either adjuvant aerosolized antibiotics plus routine IV antibiotics or aerosolized placebo plus routine IV antibiotics. Individual clinical indicators will be recorded and used to monitor the effect of aerosolized antibiotics [temperature, leukocyte count, chest radiograph appearance, ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2 ratio), mechanical ventilation status, and vital signs].

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Pulmonary Infection Score (CPIS) greater than or equal to 6
2. Intubated greater than or equal to 48 hours
3. Screened for possible eligibility
4. Bronchoscopy and bronchoalveolar lavage (BAL) or combicath performed
5. Started on empiric intravenous (IV) and inhaled antibiotics after BAL for suspected ventilator associated pneumonia (VAP)
6. > 104 Colony Forming Units (CFU) on BAL

Exclusion Criteria:

1. <18 years of age
2. Pregnant
3. Human Immunodeficiency Virus (HIV) or on chronic immunosuppressants
4. Absolute Neutrophil Count <1,000
5. Allergy to vancomycin or tobramycin
6. Anaphylaxis to penicillin
7. Cystic Fibrosis
8. Previous enrollment
9. Creatinine >2 mg/dl or doubled within the previous 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K. Bini, MD, Principal Investigator — Wright State University; Priti Parikh, PhD, Study Director — Wright State University
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klastersky J, Huysmans E, Weerts D, Hensgens C, Daneau D. Endotracheally administered gentamicin for the prevention of infections of the respiratory tract in patients with tracheostomy: a double-blind study. Chest. 1974 Jun;65(6):650-4. doi: 10.1378/chest.65.6.650. No abstract available. PMID 4208908
- [Background] Hallal A, Cohn SM, Namias N, Habib F, Baracco G, Manning RJ, Crookes B, Schulman CI. Aerosolized tobramycin in the treatment of ventilator-associated pneumonia: a pilot study. Surg Infect (Larchmt). 2007 Feb;8(1):73-82. doi: 10.1089/sur.2006.051. PMID 17381399
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] MacIntyre NR, Rubin BK. Respiratory therapies in the critical care setting. Should aerosolized antibiotics be administered to prevent or treat ventilator-associated pneumonia in patients who do not have cystic fibrosis? Respir Care. 2007 Apr;52(4):416-21; discussion 421-2. PMID 17417976
- [Background] Drew RH, Dodds Ashley E, Benjamin DK Jr, Duane Davis R, Palmer SM, Perfect JR. Comparative safety of amphotericin B lipid complex and amphotericin B deoxycholate as aerosolized antifungal prophylaxis in lung-transplant recipients. Transplantation. 2004 Jan 27;77(2):232-7. doi: 10.1097/01.TP.0000101516.08327.A9. PMID 14742987
- [Background] Wood GC, Boucher BA. Aerosolized antimicrobial therapy in acutely ill patients. Pharmacotherapy. 2000 Feb;20(2):166-81. doi: 10.1592/phco.20.3.166.34783. PMID 10678295
- [Background] Drobnic ME, Sune P, Montoro JB, Ferrer A, Orriols R. Inhaled tobramycin in non-cystic fibrosis patients with bronchiectasis and chronic bronchial infection with Pseudomonas aeruginosa. Ann Pharmacother. 2005 Jan;39(1):39-44. doi: 10.1345/aph.1E099. Epub 2004 Nov 23. PMID 15562142
- [Background] Palmer LB, Smaldone GC, Chen JJ, Baram D, Duan T, Monteforte M, Varela M, Tempone AK, O'Riordan T, Daroowalla F, Richman P. Aerosolized antibiotics and ventilator-associated tracheobronchitis in the intensive care unit. Crit Care Med. 2008 Jul;36(7):2008-13. doi: 10.1097/CCM.0b013e31817c0f9e. PMID 18552684
- [Background] Ioannidou E, Siempos II, Falagas ME. Administration of antimicrobials via the respiratory tract for the treatment of patients with nosocomial pneumonia: a meta-analysis. J Antimicrob Chemother. 2007 Dec;60(6):1216-26. doi: 10.1093/jac/dkm385. Epub 2007 Oct 13. PMID 17934205
- [Background] Claridge JA, Edwards NM, Swanson J, Fabian TC, Weinberg JA, Wood C, Croce MA. Aerosolized ceftazidime prophylaxis against ventilator-associated pneumonia in high-risk trauma patients: results of a double-blind randomized study. Surg Infect (Larchmt). 2007 Feb;8(1):83-90. doi: 10.1089/sur.2006.042. PMID 17381400
- [Background] Klepser ME. Role of nebulized antibiotics for the treatment of respiratory infections. Curr Opin Infect Dis. 2004 Apr;17(2):109-12. doi: 10.1097/00001432-200404000-00007. PMID 15021049
- [Background] Palmer LB, Smaldone GC, Simon SR, O'Riordan TG, Cuccia A. Aerosolized antibiotics in mechanically ventilated patients: delivery and response. Crit Care Med. 1998 Jan;26(1):31-9. doi: 10.1097/00003246-199801000-00013. PMID 9428540
- [Background] Smaldone GC. Advances in aerosols: adult respiratory disease. J Aerosol Med. 2006 Spring;19(1):36-46. doi: 10.1089/jam.2006.19.36. PMID 16551213
- [Background] Crowther Labiris NR, Holbrook AM, Chrystyn H, Macleod SM, Newhouse MT. Dry powder versus intravenous and nebulized gentamicin in cystic fibrosis and bronchiectasis. A pilot study. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1711-6. doi: 10.1164/ajrccm.160.5.9810080. PMID 10556145
- [Background] Heinzl B, Eber E, Oberwaldner B, Haas G, Zach MS. Effects of inhaled gentamicin prophylaxis on acquisition of Pseudomonas aeruginosa in children with cystic fibrosis: a pilot study. Pediatr Pulmonol. 2002 Jan;33(1):32-7. doi: 10.1002/ppul.10019. PMID 11747258
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Background] Pugin J, Auckenthaler R, Mili N, Janssens JP, Lew PD, Suter PM. Diagnosis of ventilator-associated pneumonia by bacteriologic analysis of bronchoscopic and nonbronchoscopic "blind" bronchoalveolar lavage fluid. Am Rev Respir Dis. 1991 May;143(5 Pt 1):1121-9. doi: 10.1164/ajrccm/143.5_Pt_1.1121. PMID 2024824

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerosolized Tobramycin or Vancomycin: Aerosolized tobramycin 300 mg diluted in 5 mL 0.9% normal saline q.12h. Aerosolized vancomycin 125 mg diluted in 5 mL 0.9% normal saline q.8h.
  Aerosolized Tobramycin or Vancomycin: Tobramycin: 300 mg diluted in 5 mL of 0.9% normal saline q.12h.
  Vancomycin: 125 mg diluted in 5 mL 0.9% normal saline q.8h.
Period: Overall Study
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Customized [Count of Participants; unit: Participants]
  Age: Under 18 | 0 | 0 | 0
  Age: Over 18 | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 3 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Patients who required ≥48 hours of mechanical ventilation [Count of Participants; unit: Participants] | 10 | 6 | 16
Patients who had a Clinical Pulmonary Infection Score ≥6. [Count of Participants; unit: Participants] — Clinical Pulmonary Infection Score is based on temperature, blood leukocytes, tracheal secretions, oxygenation, pulmonary radiography, progression of pulmonary infiltrate, and culture results. It ranges from 0-14. A total score of greater or equal to 6 is considered suggestive of pneumonia.
  Participants | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Pneumonia
Description: Recurrence after a second bronchoalveolar lavage (BAL) reveals at least one bacterial species growing at concentrations of greater than 10 to the fourth power organisms during the time period of 9-21 days after initiating therapy.
Time Frame: 9-21 days after initiating antibiotic therapy
Population: Data was not collected.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Persistence of Pneumonia
Description: Persistence will be defined as the need to continue antibiotic therapy for greater than 7 days. This is reported as the number of participants with persistence of pneumonia.
Time Frame: 8 days after initiation of therapy for pneumonia
Population: data were not collected
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Ventilator-free Days
Description: number of days not on vent in first 28 days after randomization
Time Frame: 28 days
Population: Data was not collected. Technical problems with measurement leading to unreliable or uninterpretable data.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Intensive Care Unit (ICU) -Free Days in 28 Days
Description: number of days not in ICU after initiation of therapy
Time Frame: 28 days
Population: Data not collected
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 28-day ICU Mortality
Description: number of patients treated in each arm who die in ICU within 28 days of initiation of therapy
Time Frame: 28 days
Population: Data not collected.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Renal Insufficiency
Description: patients who develop acute kidney injury after randomization
Time Frame: 28 days
Population: Technical problems with measurement leading to unreliable or uninterpretable data.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Multiple Organ Dysfunction Score Calculated at Randomization and on Day 7 of Treatment
Description: multiple organ dysfunction score at randomization and on day 7 of aerosolized antibiotics/placebo treatment
Time Frame: 7 days
Population: Data not collected. Technical problems with measurement leading to unreliable or uninterpretable data.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Emergence of Resistant Organisms
Description: patients with failure of therapy or persistence who grow resistant organisms after being treated initially
Time Frame: 28 days
Population: Data not collected. Technical problems with measurement leading to unreliable or uninterpretable data.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Antibiotic Days
Description: total days antibiotics administered for pneumonia after randomization
Time Frame: 28 days
Population: Data not collected. Technical problems with measurement leading to unreliable or uninterpretable data.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Current IRB protocol contains an erroneous exclusion criteria "Cervical spine injury with neurological deficit". Consequently and inadvertently, two subjects (002 & 011) were screened with cervical injuries and neurological deficits but screen failed out and never enrolled. One subject 004 did enroll but we have documented on the physical exam that the patient had cervical spine injury with "no neurological deficits appreciate" which permits inclusion.
Arm/Group | Aerosolized Placebo | Aerosolized Tobramycin or Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Placebo (N=10) | Aerosolized Tobramycin or Vancomycin (N=6)
Serious (Nervous system disorders) | 1 (1) | 0 (0) — Protocol has an erroneous exclusion criteria "Cervical spine injury with neurological deficit. 2 subjects were screened but screen failed out and never enrolled. 1 did enroll but has documented on the physical exam a cervical spine injury.

LIMITATIONS AND CAVEATS:
Data was not collected for the Secondary Outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT02478710/Prot_000.pdf
  • Informed Consent Form (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02478710/ICF_001.pdf